CLINICAL TRIAL: NCT04298645
Title: Controlled Nutrition Trial on the Glycaemic Response to Morning and Evening Meals With High Glycemic Index Carbohydrates Among Students With Early and Late Chronotypes-The ChroNu Study
Brief Title: Nutrition Trial on the Glycaemic Response to High GI Meals Consumed at Morning vs. Evening-The ChroNu Study
Acronym: ChroNu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paderborn University (Other)
Collaborators: German Research Foundation (Other); German Diabetes Center (Other); University of Bergen (Other)
Responsible Party: Principal Investigator, Anette Buyken, Prof. Dr. Anette Buyken, Public Health Nutrition, Paderborn University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BU1807/3-2
Record Dates: First submitted 2020-01-22; First posted 2020-03-06 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: chronotype; social jetlag; glycaemic response; glycaemic index; continuous glucose monitoring; body composition

STUDY DESIGN:
Intervention Model Description: 60 participants will be invited of which 20 participants with an earlier and 20 participants with a later chronotype are expected to finish the study. Participants will consume a meal rich in carbohydrates with a high GI on two separate days at different times. Hence, participants are randomly assigned to one group stratified by chronotype: intake of a meal with a high GI on day 5 either in the morning or in the evening. On day 7, meal timing of the high GI meal is switched. Following a 3 - day observational part on "free days", the controlled nutrition trial will last 4 days: run - in (day 4), high GI meal for breakfast/dinner (days 5 / 7), and wash - out (day 6). The trial is a two-arm cross-over study in which each participant serves as his / her own control to account for inter-individual variations in diurnal glycaemic responses.
Masking Description: Masking to the study arm is not possible for participants since the study involves consumption of "real food" to which the participants cannot be blinded. Similarly, the researchers cannot be blinded to the food provided to the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High GI carbs breakfast / dinner (Experimental): Participants will receive a meal rich in high GI carbohydrates for breakfast (day 5) first. After the wash-out day (day 6), the identical meal will be provided for dinner (day 7).
  Interventions: Other: Glycaemic response to high GI carbohydrates consumed at morning versus evening meals.
- High GI carbs dinner / breakfast (Experimental): Participants will receive a meal rich in high GI carbohydrates for dinner (day 5) first. After the wash-out day (day 6), the same meal will be provided for breakfast (day 7).
  Interventions: Other: Glycaemic response to high GI carbohydrates consumed at morning versus evening meals.

INTERVENTIONS:
Other: Glycaemic response to high GI carbohydrates consumed at morning versus evening meals. — Controlled nutrition trial on the glycaemic response to morning and evening meals with high glycemic index carbohydrates among students with early and late chronotypes.

SUMMARY:
Several studies suggest that meal timing plays an important role in the development of obesity and metabolic diseases. Especially in the evening, a high consumption of carbohydrates, which greatly increase blood glucose levels (i.e. unfavourable carbohydrates with a higher glycaemic index (GI)), has been found to adversely affect glycaemic response. However, avoidance of (unfavourable) carbohydrate consumption appears to be particularly problematic for young adults due to its interference with the timing of social life and their chronotype. The chronotype describes individual differences in sleep timing on free days and is most delayed around the age of 20. Young adults are thus prone to be exposed to a dietary misalignment when socially determined schedules, such as early lectures at universities, collide with their biologically determined later chronotype.

Therefore, it is hypothesized that dietary misalignment among young adults has detrimental short-term effects on the glucose metabolism.

In this nutrition trial, dietary misalignment is induced by providing the same meal rich in carbohydrates with a high glycaemic index (GI) on two separate days at different times: breakfast at 7:00 is assumed to reflect a schedule potentially inducing dietary misalignment among later chronotypes. Vice versa, providing this meal at dinner (20:00) may cause dietary misalignment among earlier chronotypes.

Adverse glycaemic responses are expected when the high GI meal is consumed at a time which is deviating from the schedule of the individual chronotype. A regular increase in postprandial glycaemia due to constant dietary misalignment may be important in the development of metabolic diseases.

DETAILED DESCRIPTION:
To address the hypothesis that dietary misalignment among young adults has detrimental short-term effects on glucose metabolism, participants will consume a meal rich in high GI carbohydrates on two separate days either at breakfast (7:00) or at dinner (20:00). Glycaemic responses will be monitored by a continuous glucose monitoring device (CGM) (G6, Dexcom, Inc., San Diego, CA). The CGM electrochemically measures subcutaneous interstitial glucose concentrations of each participant during the whole study. A blood glucose meter will be used to verify the functionality of the CGM (CONTOUR®NEXT ONE).

The caloric content of the meals will be tailored to the energy needs of the participants based on their age, sex and anthropometric measurements. Participants will be requested to consume the meals without any break. During the controlled nutrition trial, participants will be asked to abstain from alcohol consumption and heavy exercise and not consume any food in addition to that provided or drinks that should be explicitly avoided.

To objectively corroborate their chronotype participants will be asked to wear an accelerometer (E4 wristband, Empatica) attached to the wrist during the controlled nutrition trial. Moreover, participants are asked to record their bed times, meal timings, daily routines, and physical activities during the trial. On day 1 and day 8, anthropometric measurements will be performed to compare the body composition (Bioimpedance Analysis, SECA mBCA) before and after the controlled nutrition trial. On day 4, fasting blood samples will be collected. Before the controlled nutrition trial will start, questionnaires on daily routines, food frequency, and chronotype will be carried out.

The chronotype is defined as mid-sleep point and assessed by the Munich Chronotype Questionnaire, which is a validated questionnaire. Earlier and later chronotypes will be defined as 20% of the participants with each the earliest and later mid-sleep points among the participants of the ChroNu cohort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy students of Paderborn University
* 18 - 25 years old at time of screening for the ChroNu cohort
* 18,5 kg/m² < BMI > 30 kg/m²
* Free of diseases requiring constant or chronic medical treatment (except for oral contraceptives)
* Willingness to participate in the nutrition trial (8 days) including invasive measurements
* Fluent knowledge of the German language

Exclusion Criteria:

* students studying nutrition science at the University Paderborn
* regular smokers
* pregnancy or lactation
* chronic diseases: diabetes mellitus (all types), pre-diabetes, individuals with bleeding disorders (thrombocytopenia, haemophilia)
* contact dermatitis to adhesive plaster or skin disease that prevents the participant from wearing the CGM
* intake of medication which influence the chronotype: such as antidepressants or sleeping pills
* shift work in the past 3 months
* crossing of > 1-time zone in the past 3 months
* strict vegetarians /vegans
* individuals having an allergy or intolerance to food that is included in the diet

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Differences in the 2-h pp glycaemic response between the high GI carbohydrate meal consumed for breakfast (7:00) and the high GI carbohydrate meal consumed for dinner (20:00). | 2 hour postprandial after test meals
  2 hour post prandial response (iAUC) is calculated as the incremental area under the curve of measurements taken within the two hours after the test meals.
Differences in the 2-h pp glycaemic variability between the high GI carbohydrate meal consumed for breakfast (7:00) and the high GI carbohydrate meal consumed for dinner (20:00). | 2 hours postprandial after test meals
  the 2-h pp glycaemic variability (MAGE) is calculated as the mean amplitude of glycaemic excursions during the two hours after the test meals, i.e. both resemble summary measures calculated from repeated measurements taken the 2 h pp.

SECONDARY OUTCOMES:
Diurnal differences in the glycaemic response (iAUC) and in response to the high GI carbohydrates for dinner and the high GI carbohydrates for breakfast. | 24 hours after test meals
  24 hour post prandial response (iAUC) is calculated as the incremental area under the curve of measurements taken within the 24 hours after the test meals.
Diurnal differences in the glycaemic variability (MAGE) in response to the high GI carbohydrates for dinner and the high GI carbohydrates for breakfast. | 24 hours after test meals
  24-h pp glycaemic variability (MAGE) is calculated as the mean amplitude of glycaemic excursions during the 24 hours after the test meals, i.e. both resemble summary measures calculated from repeated measurements taken the 24 h pp.

OTHER OUTCOMES:
Blood lipids, inflammation marker, and glucose homeostasis | 7:30 on run-in day
  Blood lipids, markers of chronic inflammation, and glucose homeostasis will be measured from serum or plasma obtained from fasting whole blood samples.
  * total cholesterol (mmol/L)
  * triglycerides (mmol/L)
  * LDL- cholesterol (mmol/L)
  * HDL- cholesterol (mmol/L
  * small-dense LDL (mmol/L)
  * small-dense HDL (mmol/L)
  * high-sensitivity C-reactive protein (mmol/L)
  * Fasting blood glucose (mmol/L)
Insulin level | 7:30 run-in day
  - fasting plasma insulin level (µE/mL)
Liver enzymes | 7:30 run-in day
  * Alanine transaminase (U/L)
  * γ- Glutamyltransferase (U/L)
Clock gene expression | 7:30 run-in day
Sleep timing | 8 days
  Sleep timing (unit) will be determined using an accelerometer (Empatica E4) and manually kept diary during the 8 days of nutrition trial. This information will serve to to corroborate the chronotype of the participants.
Change in fat mass | at baseline (day 1) and after intervention (day 8)
  Body composition is electronically analyzed using Bioimpedance Analysis (BIA) (mBCA 515, SECA).
Change in Body Mass Index | at baseline (day 1) and after intervention (day 8)
  Body Mass Index (BMI) is calculated by weight(kg) / height(m)²). Weight and height are measured electronically.

CONTACTS AND LOCATIONS:
Overall Officials: Anette E Buyken, Prof. Dr., Principal Investigator — Paderborn University
Locations (1):
- Paderborn University, Paderborn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
In the University of Bergen (Department of Clinical Medicine, Center for Nutrition) explorative analyses will be performed so as to determine whether individuals with an early and late chronotype differ in their clock genes. Additional analyses may be performed to explore whether the clock genes are relevant for the effects of the intervention on the primary outcomes among both persons with early and late chronotypes. To this end they will be provided with pseudonymized data on:
  * Individual Chronotype (as assessed by the MCTQ)
  * Individual social jetlag
  * Anthropometric measurements
  * Gender
  * Birth year
  * meal timing and snacking
  * intake frequency of stimulants
  * Duration of being outdoors (contact time to the zeitgeber natural light)
  * Data on blood samples (lipid metabolism; glucose metabolism; inflammation marker; liver values)
  * Results for the primary outcome variables by study arm
Supporting Information: Study Protocol
Time Frame: Blood samples collected in TempusTM Blood RNA tubes will be collectively sent to Bergen when all samples are taken from the participants which will be September 2020 at the latest. Pseudonymized data will shared as long as need for the explorative analyses, which will be done in 2022.
Access Criteria: Pseudonymized data will be delivered personally to the University of Bergen. Requests on data will be reviewed by Mrs. Buyken,head of the study.

REFERENCES:
- [Derived] Stutz B, Krueger B, Goletzke J, Jankovic N, Alexy U, Herder C, Dierkes J, Berg-Beckhoff G, Jakobsmeyer R, Reinsberger C, Buyken AE. Glycemic response to meals with a high glycemic index differs between morning and evening: a randomized cross-over controlled trial among students with early or late chronotype. Eur J Nutr. 2024 Aug;63(5):1593-1604. doi: 10.1007/s00394-024-03372-4. Epub 2024 Apr 12. PMID 38605233